CLINICAL TRIAL: NCT05885568
Title: Validation of the Conditions of Transport of Biological Material by Drone Within the "Groupement Hospitalier de Territoire Somme Littoral Sud"
Brief Title: Validation of the Transport of Biological Material by Drone
Acronym: TRANS-AIRGHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de l'Arrondissement de Montreuil-sur-mer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0031
Record Dates: First submitted 2023-05-09; First posted 2023-06-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Drone Transport; Biological Samples; Unmanned Aerial System
Keywords: drone transport; biological samples; unmanned aerial system; UAS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- car transportation (Active Comparator): blood sample tube will be transported by courier (reference treatment)
  Interventions: Biological: blood sampling; Other: car transportation
- drone transportation (Experimental): blood sample tube will be prepared for transport by drone (departure from CHAM, 1 hour flight, arrival at CHUAP)
  Interventions: Biological: blood sampling; Other: drone transportation

INTERVENTIONS:
Biological: blood sampling — Blood sampling from healthy volunteers
Other: drone transportation — drone transportation
  Arms: drone transportation
Other: car transportation — car transportation
  Arms: car transportation

SUMMARY:
The Hospital Group of Territory Somme Littoral Sud, through its biology sector and in partnership with the company DELIVRONE, aims to engage in the experiment of transporting biological samples by means of a drone platform. Transport by air will be between the CHAM, the Abbeville Hospital and the CHU Amiens-Picardie by flying as much as possible over the waterways via the Somme. With a flight speed of around 100km/h at an altitude between 80 and 120 m, drones will be able to connect sites in less than an hour by transporting packages between 2 and 3 kg. Powered by propellers connected to rechargeable batteries, these drones do not emit CO2. This type of transport has not been validated in France by measuring the analytical impact of transport constraints for medical biology, and has never been evaluated according to the criteria of ISO 15189 standard allowing the certification of medical biology laboratories. Validation steps of this transportation method are therefore necessary on pathological samples prior to routine use.

The aim of the project is to validate the transport of biological samples by drone under defined flight conditions between CHAM and CHU Amiens-Picardie

ELIGIBILITY:
Inclusion Criteria:

* participants of legal age
* No contraindication to blood collection
* Voluntary
* informed and consenting participants

Exclusion Criteria:

* Impossible to collect sufficient blood volume
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Variation of destination arrival between both transportation types | one hour
  Arrival of the load at its destination
Variation of sample temperature during transportation | one hour
  maintaining the defined temperatures
Variation of sample allotted time after both transportation types | one hour
  Absence of variation of the allotted time of both samples after transportation
Variation of sample degradation after both transportation types | one hour
  Absence of physical degradation of both samples after transportation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No